CLINICAL TRIAL: NCT01482702
Title: Impact of Weight Loss Interventions for Overweight Breast Cancer Survivors
Acronym: VCC0910
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Kim Dittus, MD, PhD, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-031
Record Dates: First submitted 2010-04-12; First posted 2011-11-30 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Overweight; Postmenopausal; Breast Cancer
Keywords: breast cancer survivor; weight loss; postmenopausal; Weight loss for overweight postmenopausal breast cancer survivors
MeSH Terms: conditions — Overweight; Breast Neoplasms; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- weight loss intervention (Experimental): Behavioral weight loss intervention
  Interventions: Behavioral: weight loss intervention
- Weight Loss plus Resistance Training (Experimental): Behavioral weight loss intervention with the addition of resistance training
  Interventions: Behavioral: Weight Loss
- Comparator (Active Comparator): Group of women who did not receive chemotherapy
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: weight loss intervention — Behavioral weight loss intervention
  Arms: weight loss intervention
Behavioral: Weight Loss — Behavioral weight loss intervention
  Arms: Weight Loss plus Resistance Training
Behavioral: Weight Loss — Behavioral weight loss intervention
  Arms: Comparator

SUMMARY:
Obesity is an epidemic and the majority of breast cancer survivors are overweight or obese. The American Cancer Society has called for weight loss treatment to be standard of care for overweight women with breast cancer. During therapy women with breast cancer often gain weight and lose lean muscle mass. Overweight breast cancer survivors are more likely to have their cancer come back. The reason why overweight breast cancer survivors are more likely to re-occur has not been well studied, but changes in how insulin works may contribute. Overweight survivors are also at risk for the other chronic diseases associated with obesity. Fortunately, weight losses of as little as 5-7% of baseline body weight can improve risk of chronic disease. An effective behaviorally-based, lifestyle intervention delivered via the internet has been developed at the University of Vermont. This successful intervention has not been tested among breast cancer survivors. Given that women tend to lose muscle mass during cancer therapy the addition of a resistance training component to the weight loss intervention may be important. Therefore the overall goal of this project is to pilot test a proven distantly- delivered behavioral weight loss intervention among overweight breast cancer survivors and to evaluate whether a resistance program results in improvements in lean body mass, while studying how both interventions change insulin sensitivity.

Specifically, this project is a randomized, controlled clinical trial designed to test the effectiveness and acceptability of a 6-month behavioral weight loss intervention with and without resistance training. Participants will be randomized to one of two groups: 1) behavioral weight control treatment via the Internet; or 2) behavioral weight control treatment via the Internet plus a resistance training program. Women eligible to participate include overweight breast cancer survivors who are age 50 or older and 6-36 months past receiving chemotherapy. Assessments will be conducted at baseline and six months and will include measures of body weight, muscle mass, adherence to treatment, and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal (last period 12 mos prior to study enrollment or oophorectomy)
* Age 40-65
* DCIS, Stage I, II, III Breast Cancer
* BMI between 27-50
* Completed chemotherapy to treat early stage breast cancer (Stage I-III) no less then 6 months and no more than 48 months from start of study or for specific aim 3 Diagnosis of DCIS or Stage I breast cancer who did not receive chemotherapy.

Exclusion Criteria:

* Participant can not have a psychotic or central nervous system impairment that would limit compliance with study requirements
* Evidence of metastatic disease
* Chemotherapy for cancer other than breast cancer
* Diabetes mellitus, uncontrolled hypo or hyper thyroidism, liver failure
* Celiac sprue, inflammatory bowel disease
* Inability to walk for exercise
* Lymphedema as indicated by a 2 cm circumference difference at the elbow
* weight loss in the previous 6 months of 10 lbs or greater

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Identify changes in energy balance and insulin sensitivity parameters in overweight breast cancer survivors after a behavioral weight loss intervention. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Primary outcome measures include weight, fat free mass, fat mass, total and active energy expenditure, calorie intake and oral glucose tolence test
Determine whether the addition of resistance training to a behavioral weight loss intervention preserves muscle mass and improves weight loss or insulin sensitivity in breast cancer survivors. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Outcomes include weight, fat free mass, fat mass, strength (upper extremity and lower extremity) and oral glucose tolerence test

SECONDARY OUTCOMES:
Identify differences in weight loss and energy balance between post menopausal breast cancer survivors who received chemotherapy and those who did not receive chemotherapy as part of their oncologic management. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Outcomes: weight, fat mass, Fat free mass, total and active energy expenditure, calorie intake
Determine differences in insulin sensitivity parameters between post menopausal breast cancer survivors who received chemotherapy and those who did not. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Oral glusoe tolerence test
Determine feasibility, acceptability, and safety of weight loss intervention without resistance training for breast cancer survivors. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Outcomes include compliance as determined by percent of indiviudals completing each lesson and completing the program. Saftery is assessed by identifying injury or worsening lymphedema. Acceptability is determined with a survey.
Assess changes in health-related quality of life after a weight loss intervention. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Outcomes include SF-36 and FACT-fatigue surveys
Determine feasibility, acceptability, and safety of weight loss intervention with resistance training for breast cancer survivors. | Time frame is before & after the intervention. The intervention is 6 months. 4 groups of 10-22 women go through together. The groups start at different times. The last group starts May 2011. The last measurements will be obtained early Dec. of 2011.
  Outcomes include compliance as determined by percent of indiviudals completing each lesson and completing the program. Saftery is assessed by identifying injury or worsening lymphedema. Acceptability is determined with a survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Dittus, MD, PhD, Principal Investigator — University of Vermont/ Fletcher Allen Health Care
Locations (1):
- Vermont Cancer Center, Burlington, Vermont, United States

REFERENCES:
- [Derived] Dittus KL, Harvey JR, Bunn JY, Kokinda ND, Wilson KM, Priest J, Pratley RE. Impact of a behaviorally-based weight loss intervention on parameters of insulin resistance in breast cancer survivors. BMC Cancer. 2018 Mar 27;18(1):351. doi: 10.1186/s12885-018-4272-2. PMID 29587682
- See also: Vermont Cancer Center — http://vermontcancer.org